CLINICAL TRIAL: NCT06460870
Title: Effect of Mojzisova Method on Pain, Menstrual Symptom and Insomnia in Primary Dysmenorrhea
Brief Title: Effect of Mojzisova Method on Pain, Menstrual Symptom and Insomnia in PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0562 Zainab Waheed
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Primary Dysmenorrhea
Keywords: insomnia; menstrual symptom; pain; primary dysmenorrhea; stretching
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mojzisova method (Experimental): Mobilization of rib, lumbar spine, SI joint and internal rectal work. Stretching and strengthening exercises of pelvic floor, lumbar spine, sacrum and coccyx.
  Interventions: Other: Mojzisova method
- Stretching exercises (Active Comparator): Stretching exercises cobra pose, child pose and cat/cow pose.
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Other: Mojzisova method — The home based regular exercises stretching and strengthning exercises twice daily along with hot pack. Manual therapy was applied in the first half of the menstrual cycle, once a month, for one hour. It includes mobilization of ribs, lumbar spine, and sacroiliac joints as well as coccygeal treatment, and internal rectal work. The patient was received 2 sessions per month for 3 months, for 45 minutes.
  Arms: Mojzisova method
Other: Stretching exercises — Stretching exercises was performed such as cobra pose, cat/cow pose and baby pose along with hotpack for 2 sessions per month for 45 min for 3 months.
  Arms: Stretching exercises

SUMMARY:
This project was a Randomized controlled trial conducted to check the effectiveness of mojzisova method in primary dysmenorrhea for pain, menstrual symptoms and insomnia. Duration was of 6 months, convenient sampling was done, subject following eligibility criteria from DHQ hospital Toba Tek were randomly assigned, baseline assessment was done, Group A paarticipants were given baseline treatment along with mojzisova method, Group B participants were given baseline treatment along with stretching exercises, post intervention assessment was done, via WALIDD, Numeric pain rating scale (NPRS) and Pittsburgh sleep quality index (PSQI) questionnaire 45 minutes per session, 2 sessions per month for 3 months, data was analyzed by using SPSS version 26.

DETAILED DESCRIPTION:
Primary dysmenorrhea is most common reported problems to gynecologists and physical therapists. There is long history of using over the counter painkillers. Due to this there is high absenteeism from schools colleges and work. On the basis of symptoms primary dysmnorhea can be separated from secondary dysmenorrhea.Physical activity has long been used for relieving the pain, menstrual symptoms and improve insomnia. Previous studies also reported the effects of stretching exercises, core stabilizing exercises yoga, Pilates, aerobics on improving the pain and symptoms in primary dysmenorrhea. According to researcher knowledge there is limited evidence on mojzisova method that how this method improve the menstrual symptoms, pain and insomnia in primary dysmenorrhea. The aim of this study is to see the effects of mojzisova method on pain, menstrual symptom and insomnia in primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Pain must be recurrent (at least following three menstrual cycles).
* No history of any blood problems, such as thalassemia, folate insufficiency, or anemia due to a lack of iron. Five criteria to fulfill to be considered primary dysmenorrhea.
* Hypogastrium pain during menstruation.
* Irradiation of pain to lower back, lower limbs or lingual region.
* Inability to perform daily activity.
* The need for medical management or self-medication to control pain Nulliparous women with primary dysmenorrhea.

Exclusion Criteria:

* Female with history of any specific disease.
* Female with endocrine disorders.
* Had gone major surgery.
* Diagnosis of secondary dysmenorrhea.
* Having symptoms such as numbness and tingling sensation.

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 26 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
WALIDD | 4th week
  A scale-type survey (working ability, location, intensity, days of pain, dysmenorrhea [WaLIDD] score) was designed.)which integrated features of dysmenorrhea such as: 1) number of anatomical pain locations (no part of the body, lower abdomen, lumbar region, lower limbs, inguinal region), 2) Wong-Baker pain range (does not hurt, hurts a little, hurts a little more, hurts even more, hurts a lot, hurts a lot more), 3) number of days of pain during menstruation (0, 1-2, 3-4, ≥5), and 4) frequency of disabling pain to perform their activities (never, almost never, almost always, always).Each tool's variable provided a specific score between 0 and 3, and the final score ranged from 0 to 12 points.
NPRS | 4th week
  The numeric rating scale is similar to the VAS in that it is bounded at the left-most end with "no pain" and at the right-most end with "worst pain imaginable" (or something similar). The difference is that instead of a line without marks, numbers from 0 to 10 are spaced evenly across the page. Patients are instructed to circle the number that represents the amount of pain that they are experiencing at the time of the evaluation. A variation of this scale is the verbal numeric scale (VNS), in which patients are asked to verbally state a number between 0 and 10 that corresponds to their present pain intensity.
PSQI Questionnaire | 4th week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Seven component scores, ranging from 0 (no difficulty) to 3 (extreme difficulty), are obtained while assessing the PSQI. The global score, which ranges from 0 to 21, is calculated by adding the component scores. Poorer sleep quality is indicated by higher scores.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakeel Ur Rehman, Phd, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Toba Tek Singh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alikamali M, Mohammad-Alizadeh-Charandabi S, Maghalian M, Mirghafourvand M. The effects of vitamin E on the intensity of primary dysmenorrhea: A systematic review and meta-analysis. Clin Nutr ESPEN. 2022 Dec;52:50-59. doi: 10.1016/j.clnesp.2022.10.001. Epub 2022 Oct 9. PMID 36513486
- [Background] Wu L, Zhang J, Tang J, Fang H. The relation between body mass index and primary dysmenorrhea: A systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2022 Dec;101(12):1364-1373. doi: 10.1111/aogs.14449. Epub 2022 Sep 20. PMID 36124820
- [Background] Itani R, Soubra L, Karout S, Rahme D, Karout L, Khojah HMJ. Primary Dysmenorrhea: Pathophysiology, Diagnosis, and Treatment Updates. Korean J Fam Med. 2022 Mar;43(2):101-108. doi: 10.4082/kjfm.21.0103. Epub 2022 Mar 17. PMID 35320895
- [Background] Iwata M, Oikawa Y, Shimizu Y, Sakashita N, Shoji A, Igarashi A, Osuga Y. Efficacy of Low-Dose Estrogen-Progestins and Progestins in Japanese Women with Dysmenorrhea: A Systematic Review and Network Meta-analysis. Adv Ther. 2022 Nov;39(11):4892-4909. doi: 10.1007/s12325-022-02298-9. Epub 2022 Sep 1. PMID 36048405
- [Background] Al-Husban N, Odeh O, Dabit T, Masadeh A. The Influence of Lifestyle Variables on Primary Dysmenorrhea: A Cross-Sectional Study. Int J Womens Health. 2022 Apr 13;14:545-553. doi: 10.2147/IJWH.S338651. eCollection 2022. PMID 35444471
- [Background] Ferries-Rowe E, Corey E, Archer JS. Primary Dysmenorrhea: Diagnosis and Therapy. Obstet Gynecol. 2020 Nov;136(5):1047-1058. doi: 10.1097/AOG.0000000000004096. PMID 33030880
- [Background] McKenna KA, Fogleman CD. Dysmenorrhea. Am Fam Physician. 2021 Aug 1;104(2):164-170. PMID 34383437
- [Background] Kramp ME. Combined manual therapy techniques for the treatment of women with infertility: a case series. J Am Osteopath Assoc. 2012 Oct;112(10):680-4. PMID 23055467
- [Background] Kannan P, Chapple CM, Miller D, Claydon-Mueller L, Baxter GD. Effectiveness of a treadmill-based aerobic exercise intervention on pain, daily functioning, and quality of life in women with primary dysmenorrhea: A randomized controlled trial. Contemp Clin Trials. 2019 Jun;81:80-86. doi: 10.1016/j.cct.2019.05.004. Epub 2019 May 7. PMID 31071464
- [Background] Samy A, Zaki SS, Metwally AA, Mahmoud DSE, Elzahaby IM, Amin AH, Eissa AI, Abbas AM, Hussein AH, Talaat B, Ali AS. The Effect of Zumba Exercise on Reducing Menstrual Pain in Young Women with Primary Dysmenorrhea: A Randomized Controlled Trial. J Pediatr Adolesc Gynecol. 2019 Oct;32(5):541-545. doi: 10.1016/j.jpag.2019.06.001. Epub 2019 Jun 11. PMID 31195099